CLINICAL TRIAL: NCT06554756
Title: Annexin Levels in GCF Determine the Imbalance of Periodontal Inflammatory Regulation
Brief Title: Annexin Levels of Periodontal Inflammatory Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Melis Yilmaz, Associate Prof Dr, Medipol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 635
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases; Inflammation
Keywords: periodontal disease; annexin
MeSH Terms: conditions — Periodontal Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Saliva, serum and gingival crevicular fluid of periodontitis patients collected for analyzing anxa1, anxa2 and IL-1beta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Other): Saliva, serum and GCF collection of patients and samples molecules analysis
  Interventions: Other: Saliva, serum and GCF sampling
- Experimental (Experimental): Salivary, serum and GCF ANXA1, ANXA2 and IL-1beta observation Saliva, serum and GCF samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for ANXA1, ANXA2 and IL-1beta using commercial ELISA kits (Elabscience, Houston, Texas, USA and Bioaasay Technology Laboratory (BT-Lab), Shanghai, China, respectively) according to the manufacturer's instructions.
  Interventions: Other: Saliva, serum and GCF sampling

INTERVENTIONS:
Other: Saliva, serum and GCF sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Gingival crevicular fluid (GCF) samples were taken from the vestibular, mesial, and distal surfaces of a single-rooted tooth with standard paper strips (Periopaper, Oraflow Inc., Plainview, NY, USA). Saliva, GCF and serum were then stored at -80 °C until analysis.

SUMMARY:
ANXA1, a member of the annexin family, plays a role in the resolution of inflammation and the regulation of anti-inflammatory responses, while ANXA2 is involved in the initiation of the inflammatory responses. The aim of this study was to determine the effects of annexin family (ANXA1 and ANXA2) in periodontal disease.

DETAILED DESCRIPTION:
Healthy participants (n:25) and stage III, grade B periodontitis (n:25) patients enrolled for this study. Clinical periodontal parameters and PISA levels were noted. Serum, saliva, and GCF samples were collected to measure the ANXA1, ANXA2 and IL-1β levels.

ELIGIBILITY:
Inclusion Criteria:

systemically healthy

* clinical diagnosis of periodontitis
* clinical diagnosis of periodontal health

Exclusion Criteria:

* • history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)

  * nonsurgical periodontal treatment (previous 6 months)
  * surgical periodontal treatment (previous 12 months)
  * presence of<10 teeth
  * current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
  * diabetes
  * diagnosis of rheumatoid arthritis
  * pregnancy
  * lactating
  * smoking
  * excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 6 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 6 months
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
Saliva, serum and GCF samples processing and analyses | 1 month
  Saliva, GCF and serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for ANXA1, ANXA2 and IL-1beta using commercial ELISA kits

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz M, Bal I, Hanli S, Turkmen E, Balci N, Toygar HU. Annexin levels in GCF determine the imbalance of periodontal inflammatory regulation. Sci Rep. 2024 Nov 21;14(1):28833. doi: 10.1038/s41598-024-80418-x. PMID 39572681